CLINICAL TRIAL: NCT02341222
Title: "BP as a Super-light Mesh and as a New Fixing Device for General, Emergency and Prosthetic Surgery. The BP Implantation Effects on Immunity System, on the Metabolism and on Sealing. Preliminary Experimentation of Small Feasibility Study"
Brief Title: BP as a Super-light Mesh and as a New Fixation Device for General Surgery -DM108/2008-B
Acronym: DM108/2008-B
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Sannio (Other); P Consentino Appialab Veterinary Reseach Labaratory (Unknown); Catholic University of the Sacred Heart (Other); E D'Amore Istituto Superiore Sanità (Unknown)
Responsible Party: Principal Investigator, Massimo Chiaretti, Dr, PhD, MSc, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DM108/2008-B
Record Dates: First submitted 2014-12-15; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2014-07

CONDITIONS: Hernia
Keywords: hernia prosthetic surgery; incisional hernia prosthesis; prosthesis mesh fixation; prosthesis mesh biocompatibility
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BP self-standing felt device (Experimental): BP device will be implanted under fascia group-A, operated subjects. A lumbar 4-5 cm incision will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, with a blunt dissection the fascia will be separated from muscles. Fifteen rats will receive 2x2cm2 samples of BP (Buckypaper) in a pocket created between muscular fascia and large muscles. The rough opaque surface will face the muscle surface and the smooth brilliant surface will face the lower muscular fascia surface, without fixation with stitches. Then the scar will be sutured with absorbable stitches on the fascia incision edge and not absorbable stitches on the skin.
  Interventions: Device: BP self-standing felt device
- PR (parietene) mesh device (Active Comparator): A lumbar 4-5 cm incision will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, with a blunt dissection the fascia will be separated from muscles. Fifteen rats (hereafter defined as BPR16-BPR30) will receive 2x2cm2 samples of PP (polypropylene) in a pocket created between muscular fascia and large muscles. The polypropylene prosthesis will be fixed to the muscle with absorbable sutures surface and then the muscular fascia will be sutured over the prosthesis, with absorbable stitches on the fascia. Not absorbable stitches will be sutured on the skin.
  Interventions: Device: PR Parietene mesh device

INTERVENTIONS:
Device: BP self-standing felt device — BP device will be implanted under fascia group-A, operated subjects. A lumbar 4-5 cm incision will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, with a blunt dissection the fascia will be separated from muscles. Fifteen rats will receive 2x2cm2 samples of BP (Buckypaper) in a pocket created between muscular fascia and large muscles. The rough opaque surface will face the muscle surface and the smooth brilliant surface will face the lower muscular fascia surface, without fixation with stitches. Then the scar will be sutured with absorbable stitches on the fascia incision edge and not absorbable stitches on the skin.
  Other Names: BP (Buckypaper NanoLab Inc., Newton, MA 02458 USA); V-Loc 180 (ref VLOCL0024, lot. A1D0899)
  Arms: BP self-standing felt device
Device: PR Parietene mesh device — Fifteen rats (hereafter defined as BPR16-BPR30 B-group control subjects) will receive 2x2cm2 samples of PP (polypropylene) in a pocket created between muscular fascia and large muscles. A lumbar 4-5 cm incision will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, with a blunt dissection the fascia will be separated from muscles. Fifteen rats (hereafter defined as BPR16-BPR30) will receive 2x2cm2 samples of PP (polypropylene) in a pocket created between muscular fascia and large muscles. The polypropylene prosthesis will be fixed to the muscle with absorbable sutures surface and then the muscular fascia will be sutured over the prosthesis, with absorbable stitches on the fascia. Not absorbable stitches will be sutured on the skin.
  Other Names: PR Parietene mesh Tyco (ref. PP3030, lot. SIK00587); V-Loc 180 (ref VLOCL0024, lot. A1D0899)
  Arms: PR (parietene) mesh device

SUMMARY:
The Buckypaper (BP) is an innovative material that has attracted the attention of many research groups engaged in the study of its possible applications in various technological fields. Our purpose is demonstrate the viability of the application of nanotechnologies to the General Surgery in human with thwe use of a new self standing prosthetic device for the reconstruction of abdominal wall defects.

DETAILED DESCRIPTION:
The interesting material properties, such as good mechanical strength, electrical conductivity, low density, porosity adaptable, are closely associated to the intrinsic characteristics of carbon nanotubes (CNTs), of which BP is made . The high surface development of CNT, in addition to promoting their aggregation, allows the preparation of micro-and nano-porous membranes that exclude the passage of colloidal particles with a diameter greater than 50 nm. The micro-porous structure, also gives the BP high capacity to absorb liquids, such as water, for which the effect of capillarity, penetrates quickly in the mesh material. This could be a possible interpretation of the rapid and effective adhesion of BP to humid biological tissues observed in our preliminary studies on the effects of the BP implanted in vivo.

The bio-adhesion of BP has been documented in ex vivo preliminary experiments mechanical peeling (bench surgery). The results showed that the force required the posting of BP from organic support is much greater than that required for the conventional prosthesis made from polymer networks, commonly used in human hernia surgery fixed with fibrin glue or synthetic materials. Based on these assessments the use of BP could be introduced in the field of prosthetic surgery.

Based on these assessments and based on the potential offered by the use of BP in the field of prosthetic surgery, deductible by the intrinsic characteristics of the material in this project is expected to further research for the development of a new generation of prosthetic materials for humans use, easily implantable by the surgeon without the need for sutures, graphs and / or biological glues.

The reasons are:

1. stitches: they could tighten the knot vessels (ischemia-atrophy) or nerves (chronic pain);
2. graphs: placing blind and can cause bleeding or pain;
3. biological glues: derived from the plasma of donors and thus could transmit diseases unknown.

It is still unknown if BP has the appropriate mechanical properties to withstand the stresses that occur on the abdominal wall and In any case is documented the good bio-adhesion on living tissues and anatomical preparations, but only if made humid.

Exploiting the functional groups present or introduced into the crystalline structure of MWCNTs (multiwall carbon nanotube) and/or on the polymer, it will be possible to implant on the muscle/muscular fascia surface, the composite material, to obtain gripping. Moreover, biologically active molecules, with functions antimicrobial, anti-adhesive, anti-inflammatory or analgesic, can be introduced into the crystalline structure of MWCNTs, for modulate the inflammatory response and the incorporation of the implanted material in the fibrous scar.

We would like investigate the effects of exposition to BP fragments on healthy tissues and CaCo2 cells (Cancer Colon cluster), MCF-7 (Michigan Cancer Foundation-7), a breast cancer cell line, and hSCs (healthy smooth-muscle cells) of thyroid artery.

The objective of this project is to obtain results that can direct the search for the ultimate realization of a prosthetic device for use in human abdominal surgery.

Our Research Group proposes that the present research program has all the skills to achieve all the objectives .

The protocol have been drawn in the respect of environmental policies, and ethical principles on experimentation on animal model, in accordance with the guidelines of the European Union (86/609/EEC-European Economic Community), and the Italian Law n° 116/92.

The clinical-chemical parameters examined from blood samples of 1 ml will be: BUN (blood urea nitrogen), blood glucose, creatinine, sodium, potassium, calcium, magnesium, albumin, total Blood proteins levels, SGOT (serum glutamate oxaloacetate transaminase), SGPT (serum glutamate pyruvate transaminase), GGT (galactosylhydroxylysyl glucosyltransferase), ALP (alkaline phosphatase) and fractionated bilirubin, PT (prothrombin time), APTT/PTT (activated partial thromboplastin time / prothrombin time), Fibrinogen, CBC (complete blood count) formula, lymphocyte sub-populations, C-reactive protein, erythrocyte sedimentation rate.

This procedure will be performed under sedation and followed by body weight check and the pick-up of a blood sample. The same procedure will be repeated twice at the intervention and after 35 days at the sacrifice.

At the time of sacrifice will be prepared anatomic samples of all the viscera and of the implantation site, to be studied histologically. Pathohistological samples for microscopic examination will be prepared. Portions of BP implanted in BPR1-BPR15 will be excised with all the surrounding fascia, dermal and muscular tissues. The same procedures will be performed, also in PRR16-PRR30 group.

The post-operative pain, as in the human, it will be mild, and will be treated with analgesics according to techniques standardized in humans. In our experience, the animals undergo to prosthetic surgery, both the experimental and the control group, will treated with prophylactic antibiotics and pain medication in the immediate post -operative, and will be closely watched.

Even if in animal model, the sterility of all the surgical procedure prevents inflammation, edema and sepsis and abscesses and ensures a low level of postoperative pain. The days after the surgical procedure is expected a moderate appetite of the operated animals and mild clinical symptoms related to the post-operative .

All treated animals will be observed daily to carefully control the amount of food that will be consumed and thus the potential loss of appetite. Will be look for evidence of possible inflammatory and degenerative processes affecting the skin of the abdominal wall, the symptoms of infection or rejection of the prosthesis. If weight loss will be excessive (e.g. more than 10% of the normal weight of an animal of the same race, the same age and in comparison to the control group), or the animal will show clinical symptoms of suffering more than a normal postoperative, will be subjected to general anesthesia and then deleted.

The analgesic and antibiotic therapy performed in the postoperative period will be as follows :

Antibiotic : enrofloxacin 2.5 mg /kg /day I.M. for 5/ 7 days; and anti-inflammatory analgesic : ketoprofen, Findol 10%, 0.3 ml/10kg/die i.m. for 3 /5 days. If necessary will be given also tramadol, 2-4 mg /kg/day in the first 2 /3 days post-intervention . The surgical wound will be checked daily.

The clinical -chemical parameters examined from blood samples of 3 ml will be: BUN (Blood Urea Nitrogen), blood glucose, creatinine, sodium, potassium, calcium, magnesium, albumin, total proteinemia and Blood protein level, SGOT(Serum Glutei Oxaloacetic Transaminase), SGPT(Serum Glutamic PyruvateTransaminase), GGT(gamma glutamyl transferase), ALP(alkaline phosphatase) and fractionated bilirubin, PT(Prothrombin Time), APTT/PTT(Activated partial thromboplastin time), Fibrinogen, CBC(Complete Blood Count) formula, lymphocyte subpopulations, C-reactive protein, erythrocyte sedimentation rate.

At the sacrifice the organ samples will be fixed in 10% buffered formalin, cut and stained with Haematoxylin and Eosin (H&E) for histological observation.

ELIGIBILITY:
Inclusion Criteria: female Sprague Dawley rats of 300-500 grams of body weight

Exclusion Criteria:

* any kind of illness in rat subjects
* out breed animals

Ages: 2 Months to 4 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
bio-compatibility by liver performance (by SGOT(Serum Glutamic Oxaloacetic Transaminase) | 5 weeks
  bio-compatibility of Buckypaper implanted in a lumbar scar by evaluation of liver function by SGOT(Serum Glutamic Oxaloacetic Transaminase), SGPT(Serum Glutamic PyruvateTransaminase), GGT(gamma glutamyl transferase), ALP(alkaline phosphatase) and fractionated bilirubin, PT(Prothrombin Time), APTT/PTT(Activated partial thromboplastin time), Fibrinogen. The evaluation will be performed at the beginning of experimentation and at the sacrifice after 35 days and will be evaluated the difference (delta) before and after implantation of BP

SECONDARY OUTCOMES:
cancer cell viability if exposed to BP | 5 weeks
  We will investigate the effects of exposition to BP fragments on healthy tissues and CaCo2 cells (Cancer Colon cluster), MCF-7 (Michigan Cancer Foundation-7), a breast cancer cell line, and hSCs (healthy smooth-muscle cells) of thyroid artery.
bio-compatibility by kidney performance (by BUN and blood creatinine, and creatinine clearance) | 5 weeks
  bio-compatibility of Buckypaper implanted in a lumbar scar by evaluation of kidney by BUN and blood creatinine, and creatinine clearance. The evaluation will be performed at the beginning of experimentation and at the sacrifice after 35 days and will be evaluated the difference (delta) before and after implantation of BP
bio-compatibility by marrow biologic performance (by CBC(Complete Blood Count) | 5 weeks
  bio-compatibility of Buckypaper implanted in a lumbar scar by evaluation of marrow function by CBC(Complete Blood Count) formula, lymphocyte subpopulations, C-reactive protein, erythrocyte sedimentation rate. The evaluation will be performed at the beginning of experimentation and at the sacrifice after 35 days and will be evaluated the difference (delta) before and after implantation of BP

OTHER OUTCOMES:
bio-adhesivity in mm | 5 weeks
  bio-adhesivity of the prosthetic material by the displacement in mm of the prosthesis from the implantation site

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Chiaretti, MD, PhD, MSc, Principal Investigator — University of Roma La Sapienza
Locations (1):
- National Health Institute (ISS Istituto Superiore di Sanità), Viale Regina Elena 299, Rome, Roma, Italy

REFERENCES:
- [Result] Martinelli A, Carru GA, D'Ilario L, Caprioli F, Chiaretti M, Crisante F, Francolini I, Piozzi A. Wet adhesion of buckypaper produced from oxidized multiwalled carbon nanotubes on soft animal tissue. ACS Appl Mater Interfaces. 2013 May 22;5(10):4340-9. doi: 10.1021/am400543s. Epub 2013 May 1. PMID 23635074
- [Result] Bellucci S, Chiaretti M, Onorato P, Rossella F, Grandi MS, Galinetto P, Sacco I, Micciulla F. Micro-Raman study of the role of sterilization on carbon nanotubes for biomedical applications. Nanomedicine (Lond). 2010 Feb;5(2):209-15. doi: 10.2217/nnm.09.100. PMID 20148633
- [Result] Bellucci S, Chiaretti M, Cucina A, Carru GA, Chiaretti AI. Multiwalled carbon nanotube buckypaper: toxicology and biological effects in vitro and in vivo. Nanomedicine (Lond). 2009 Jul;4(5):531-40. doi: 10.2217/nnm.09.36. PMID 19572819
- [Result] Di Sotto A, Chiaretti M, Carru GA, Bellucci S, Mazzanti G. Multi-walled carbon nanotubes: Lack of mutagenic activity in the bacterial reverse mutation assay. Toxicol Lett. 2009 Feb 10;184(3):192-7. doi: 10.1016/j.toxlet.2008.11.007. Epub 2008 Nov 21. PMID 19063954
- [Result] Catani M, De Milito R, Spaziani E, Chiaretti M, Manili G, Capitano S, Di Filippo A, Simi M. [Laparoscopic inguinal hernia repair "IPOM" vs "open tension free". Preliminary results of a prospective randomized study]. Minerva Chir. 2003 Dec;58(6):783-9. Italian. PMID 14663405
- See also: preliminary results, doi:10.1088/0953-8984/20/47/474203 — http://iopscience.iop.org/0953-8984/20/47/474203/